CLINICAL TRIAL: NCT07212790
Title: Feasibility of REAL-Fam to Support Diabetes Self-Management, Family Participation, and Child Health
Brief Title: REAL-Fam Feasibility Study for Youth Diabetes Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Occupational Therapy Foundation (Other); Creighton University (Other); DexCom, Inc. (Industry); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-0708
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Rural Health; Occupational Therapy; Diabetes Management; Behavioral Health; Family-Centered Care; Psychosocial; Family Health; Diabetes; Behavioral Intervention; Child Health; Family Participation; Diabetes Quality of Life
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: There will be an intervention group and an attention group participating over the same 14 week study period.
Who Masked: Outcomes Assessor
Masking Description: The statistician who is performing randomization and statistical analysis of data will be blinded to which arm of the study to which a participant was selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REAL-Fam Intervention Group (Experimental): 8 caregiver-child dyads will receive the Resilient, Empowered, Active Living for Families intervention. This is an occupational therapy family coaching intervention, which will be delivered via 12 weekly telehealth sessions.
  Interventions: Behavioral: REAL-Fam Occupational Therapy Family Coaching
- Attention Group (No Intervention): 8 caregiver-child dyads will receive 3 attention group sessions with a research team member and engage in activities such as creating music play lists, playing games, and having conversation without specialized healthcare services.

INTERVENTIONS:
Behavioral: REAL-Fam Occupational Therapy Family Coaching — The REAL-Fam draws on the expertise of occupational therapy in evaluating the fit between the demands of everyday activities and the skills and abilities of the parent-child dyads. The dyad and the occupational therapist will be equipped to co-develop personalized strategies to enable participation in these meaningful occupations. It facilitates the family's consistent, habitual, and effective performance of their child's diabetes management tasks into their personalized daily routines. Emphasis is on the creation or modification of family-centered diabetes management and routines and catered to the child's developmental needs. Due to the complexity of diabetes management cares and the child's age, the caregiver will be present for all sessions. When working towards a caregiver-centered outcome, the caregiver will participate with little child involvement. When working toward a child-centered outcome, the child will be the focus of that session.
  Arms: REAL-Fam Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if the REAL-Fam occupational therapy intervention is feasible to study in a larger-scale randomized controlled trial. It will also seek to understand how the intervention influences how a rural family participates in and manages their child's type 1 diabetes, their family quality of life, and the child's health outcomes. The main questions it aims to answer are:

* Primary Aim 1: Evaluate the recruitment capability, participant inclusion criteria, assessment selection and process, and data.
* Primary Aim 2: Evaluate the participant acceptability of and interventionist fidelity to the intervention.
* Secondary Aim: Evaluate families' preliminary outcomes to the REAL-Fam on family quality of life and participation, diabetes management self-efficacy, and child blood glucose stability.

Researchers will compare the REAL-Fam intervention to the Attention Group to see if there are changes in family diabetes-related health routines and psychosocial aspects of managing a child's type 1 diabetes.

Participants will:

* Children will wear continuous glucose monitors for study period
* Caregiver participants will complete baseline and post-intervention surveys
* Intervention Group: engage in 12 audio/video telehealth sessions with REAL-Fam intervention
* Attention Group: engage in 3 audio/video Zoom meetings without specialized services
* Complete a post-study interview

DETAILED DESCRIPTION:
The prevalence of type 1 diabetes (T1D) is increasing among youth in the U.S., with higher incidence rates documented in rural communities compared to their urban peers. This rise is especially concerning for rural families, because they are at risk for healthcare disparities resulting from transportation challenges, lack of healthcare access, decreased financial stability, and other social determinants of health. The Resilient Empowered Active Living for Families (REAL-Fam) occupational therapy telehealth intervention provides a practical, immediate solution to increase access to low-cost, quality healthcare services for rural-dwelling caregivers and children living with T1D. Utilizing community-engaged research methods, this randomized clinical trial with follow-up interviews examines the feasibility of the 12-week REAL-Fam intervention group (n=8 dyads) compared to an attention group (n=8 dyads) for rural-dwelling caregiver/child dyads to improve the a) caregivers' diabetes management self-efficacy, b) caregivers' quality of life, and the c) children's glycemic levels. The REAL-Fam is innovative because it will extend diabetes care beyond glucose monitoring to include culturally sensitive healthcare experiences, family-centered behavioral interventions, healthy habit and routine training, and school and childcare participation strategies within the scope of occupational therapy. The successful evaluation of the REAL-Fam is critical to evaluate the protocol and support a full-scale clinical trial, which may inform other historically underrepresented socio-demographic groups that may not have access to ongoing diabetes healthcare services.

The findings from this study will inform healthcare practitioners, patients, and other stakeholders of the needs of rural families who are caring for a child with T1D and their urgent healthcare needs, such as improving quality of life and increasing access to specialized healthcare services. From the interdisciplinary team's past research focusing on T1D stakeholder needs in rural communities, it was apparent that many caregivers reported a need to access specialized diabetes care quicker after their child's diagnosis, which without this access they experienced poor health outcomes. Overall, successful evaluation of the REAL-Fam telehealth intervention is an important, necessary step to support future studies that may contribute to the advancement of T1D healthcare practices and improved child health outcomes for rural dwelling families.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver over 19 years old and designated guardian or parent to a child living with Type 1 Diabetes;
* Live in a rural area over 1 hour from pediatric endocrinology care team;
* Access to reliable internet

Exclusion Criteria:

* Caregiver who is not completing any supervision/support for their child's diabetes management;
* If the child is currently receiving occupational therapy services;
* Has a severe developmental, intellectual, or neurological disability

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Families Consented Versus Approached | 12-week post treatment initiation
  One feasibility measure was to evaluate the number and percentage of families consented compared to those approached for participation in the study.
Number and Percentage of Standard of Care Condition Participants Retained vs Enrolled | 12-week post treatment initiation
  Number and Percentage of standard of care condition participants retained in the study compared to those enrolled. Retention is defined as participants who completed post-intervention assessments.
Number and Percentage of Intervention Group Condition Participants Retained vs Enrolled | 12-week post treatment initiation
  Number and Percentage of Intervention Group participants retained in the study compared to those enrolled. Retention is defined as participants who completed post-intervention assessments.
Number and Percentage of Surveys Completed by Participants Who Completed the Study | 12-week post treatment initiation
  Number and Percentage of surveys over time completed by participants who completed the study.
Number and Percentage of attendance at telehealth sessions | 12-week post treatment initiation
  The total number/amount of sessions attended out of the total number of sessions available, reported as both the total number and the percentage.
Number and percentage of dyads enrolled for the different recruitment strategies | 12-week post treatment initiation
  For each recruitment strategy, the researchers will document the total number and percentage of how many families were eligible, approached, and enrolled
Telehealth Satisfaction Survey | 12-week post treatment initiation
  A self-reported questionnaire for caregivers to rate how satisfied they were with the telehealth sessions (a measure of study acceptability). It includes 10 questions with 1-4 ratings, with higher scores indicating higher levels of satisfaction.
Training Satisfaction Rating Scale | 12-week post treatment initiation
  A self-reported questionnaire for caregivers to rate their satisfaction with the REAL-Fam intervention. It includes the following subdomains: Objectives and content (3 questions); Method of training context (6 questions); Usefulness and overall rating (3 questions). Items are rated on a 1-5 scale, with higher scores indicating higher levels of acceptability.
Study Specific Interview Guide | 12-week post treatment initiation
  A semi-structured interview guide to qualitatively assess feasibility and acceptability of the REAL-Fam intervention framework. It includes questions related to recruitment and enrollment (3 questions); scheduling and time commitment (3 questions); assessments and data collection (3 questions); technology use (2 questions); overall burden/ease (2 questions); perceived value of the intervention ( 2 questions); engagement and enjoyment (2 questions); format delivery (2 questions); relevance to family's life (2 questions); therapist interaction (2 questions); rural context (2 questions); modules and content (3 questions); habit & routine focus of the intervention (3 questions); perceived changes/impact (2 questions); recommendations for improvement (2 questions); and overall reflections (2 questions). Qualitative results will be reported by each sub-domain.

SECONDARY OUTCOMES:
WHO Quality of Life, Brief (WHOQOL-BREF) | Baseline and 12-week post treatment initiation
  Self-reported quality of life; higher score = better quality of life. The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall QOL and general health. Subscales (domains): Physical Health (7 items) Psychological Health (6 items) Social Relationships (3 items) Environment (8 items) Scoring: Items scored 1-5. Raw domain score is the sum of respective item scores. All domain scores are then normalized to a range of 0-100. Results reported by each sub-domain and by total score.
Diabetes Health Management Performance Scale - Parents of Children | Baseline and 12-week post treatment initiation
  Self-reported performance in various diabetes health management tasks; higher score = higher level of performance with diabetes self management. Includes two parts to the assessment. Part A has the caregiver rate their performance in each category from the past 3 months. There are 5 subdomains: Diabetes Self-Management, (6 questions); Nutrition (2 questions); Physical Activity & Exercise (2 questions); School and Childcare (3 questions); and Lifestyle Management (12 questions). Part B has the caregiver rate their child's performance in the following subdomains: Diabetes Self-Management (5 questions); Nutrition (2 questions); Physical Activity and Exercise (2 questions); School and Childcare (1 question); and Lifestyle Management (3 questions). Results reported by each subdomain.
Problem Areas in Diabetes - Parents of Children | Baseline and 12-week post treatment initiation
  A self-reported questionnaire for caregivers to report any potential difficulties with managing their child's diabetes cares. It includes 16 questions, with a rating of 1-6, with higher scores indicating a more serious problem with managing their child's diabetes. Results reported as one total score.
Diabetes Family Conflict Scale - Revised | Baseline and 12-week post treatment initiation
  A self-reported questionnaire for caregivers to report any potential family conflicts with managing their child's diabetes' cares. It includes 19 questions, with a 1-3 rating, and higher ratings indicating more family conflict.
Self-Efficacy for Diabetes Scale (MSED) | Baseline and 12-week post treatment initiation
  A self-reported questionnaire for caregivers to report their confidence with managing their child's diabetes self-cares. Includes 17 questions, on a 1-5 rating, with higher scores indicating higher levels of confidence in completing diabetes self management.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jewell, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill